CLINICAL TRIAL: NCT01590784
Title: The Reliability and Validity of the Thai Version of Calgary Depression Scale for Schizophrenia (CDSS)
Brief Title: Reliability and Validity of Thai Calgary Depression Scale of Schizophrenia (CDSS)
Status: Completed | Type: Observational
Sponsor: Chiang Mai University (Other)
Responsible Party: Principal Investigator, Sirijit Suttajit, University instructor, Chiang Mai University
Other Study IDs: PSY-11-09-09-12
Record Dates: First submitted 2012-04-27; First posted 2012-05-03 (Estimated); Last update posted 2016-07-28 (Estimated); Status verified 2016-07

CONDITIONS: Depression
Keywords: Depression; Schizophrenia
MeSH Terms: conditions — Depression; Schizophrenia

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
Depression in patients with schizophrenia is common. Several factors was found to be associated with depression including medical illness, quality of life, positive symptoms, and typical antipsychotics. The Calgary depression scale of schizophrenia (CDSS) is commonly used for screening depression in schizophrenia,however; the Thai version of CDSS has not been validated.

This study aims to a.) test the reliability and validity of the Thai version of Calgary depression scale of schizophrenia (CDSS) and b.) identify the prevalence and factors associated with depression in patients with schizophrenia including quality of life, type of antipsychotic drugs, and severity of schizophrenia in 60 patients with schizophrenia at the Faculty of Medicine, Chiang Mai University, Thailand.

DETAILED DESCRIPTION:
Measurements:

The Thai version of Calgary depression scale of schizophrenia (CDSS), Positive and Negative Syndrome Scale (PANSS), Hamilton Rating Scale for Depression-17 (HAM-D 17), Montgomery-Asberg Depression Rating Scale (MADRS), the Thai abbreviated version of World Health Organization quality of life (WHOQOL-BREF-THAI).

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or over
* Diagnosis of schizophrenia according to DSM-IV-TR

Exclusion Criteria:

* Having organic brain syndrome
* Not fluent in Thai

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pariticipants diagnosed with schizophrenia according to DSM-IV-TR.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2012-01; Primary Completion 2014-06 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
The reliability of the Thai version of the Calgary Depression Scale for Schizophrenia (CDSS) in schizophrenia patients. | 3 months
  The inter-rater reliability, the test-retest reliability will be analyzed.
The validity of the Thai version of the Calgary Depression Scale for Schizophrenia (CDSS) in schizophrenia patients. | 3 months
  The Positive and Negative Syndrome Scale (PANSS), Hamilton Rating Scale for Depression-17 (HAM-D 17), Montgomery-Åsberg Depression Rating Scale (MADRS) will be administered by the first rater, whereas the CDSS will be assessed by a second independent rater.

SECONDARY OUTCOMES:
The prevalence of depression in patients with schizophrenia | 3 months
  The point prevalence of depression in patients with schizophrenia will be presented in percentage.
The association between depression in schizophrenia and quality of life. | 3 months
  The association between depression in schizophrenia and quality of life (WHOQOL-BREF-THAI).
The association between depression in schizophrenia and type of antipsychotic drugs. | 3 months
  The association between depression in schizophrenia and type of antipsychotic drugs (typical vs atypical).
The association between depression in schizophrenia and severity of schizophrenia. | 3 months
  The association between depression in schizophrenia and severity of schizophrenia (PANSS score).

CONTACTS AND LOCATIONS:
Overall Officials: Sirijit Suttajit, MD, MSc, Study Director — Chiang Mai University
Locations (1):
- Chiang Mai University, Chiang Mai, Chiang Mai, Thailand